CLINICAL TRIAL: NCT06180603
Title: Strategy for Prompt and Effective Thoracentesis in the Emergency Department: A Multicenter Randomized Clinical Trial
Brief Title: Strategy for Prompt and Effective Thoracentesis in the Emergency Department
Acronym: SPEEDTAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU307272
Record Dates: First submitted 2023-11-09; First posted 2023-12-22 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pleural Effusion; Pleural Diseases; Heart Failure
Keywords: Thoracentesis; Emergency department; Treatment methods
MeSH Terms: conditions — Pleural Effusion; Pleural Diseases; Heart Failure; Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard of care thoracentesis in the radiology department ( passively drainage using gravity)
  Interventions: Procedure: Gravity fluid drainage in the radiology department
- Intervention group (Experimental): Thoracentesis in the emergency department (manual fluid drainage using a syringe connected to a three-way stopcock)
  Interventions: Procedure: Manual drainage in the emergency department

INTERVENTIONS:
Procedure: Gravity fluid drainage in the radiology department — Patients will be referred to the radiology department. Thoracentesis will be performed according to local guidelines.
  Arms: Control group
Procedure: Manual drainage in the emergency department — Thoracentesis will be performed according to current guidelines in the emergency department. Fluid will manually be drained using a syringe connected to a three-way stopcock. Thoracentesis will be stopped early if:
  Arms: Intervention group

SUMMARY:
The SPEEDTAP-trial is a prospective, randomised, investigator-initiated, multicenter, clinical superior trial investigating two thoracentesis methods in four emergency departments (ED) in Central Denmark Region. Patients are randomised to either manual fluid removal in the ED or passively fluid drainage using gravity in the radiology department (standard of care). Primary outcome: time from clinical indication to complete drainage and 188 patients will be included. Key secondary outcomes include length of stay, ED admission to ED discharge and safety end-points.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years admitted to the ED
* Pleural effusion detected by any imaging modality (e.g., bedside ultrasound, chest x-ray, computed tomography)
* Clinically justified need for thoracentesis ( symptomatic relief and/or define the etiology of the effusion
* Without contraindication for thoracentesis in the emergency department (e.g., anticoagulant treatment)

Exclusion Criteria:

* Life-threatening respiratory distress
* Not able to give consent
* Previous pleurodesis
* Effusion does not appear free-flowing due to septations or loculations / suspected empyema
* Prior enrollment in the trial
* If randomization is not possible because decision to insert a pigtail catheter is made in the radiology department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from identification of the clinical indication for thoracentesis to complete drainage | From date and time for randomization until the date and time removal of catheter, assessed up to 3 month
  Time from identification of the clinical indication for thoracentesis is defined as the time patient is randomized. The time of complete drainage is defined by removal of pigtail catheter

SECONDARY OUTCOMES:
Hospital length of stay (days) | Date of admission until date of hospital discharge, assessed up until 3 month
  Defined as from date of admission until the date of hospital discharge
Duration of procedure (time) | from date and time for insertion until date and time for removal, assessed up until 3 month
  Defined as from date and time for insertion of catheter until date and time for removal of catheter
Patients degree of chest discomfort (score) | from date of indication until removal of catheter, assessed up until 3 month
  Chest discomfort will be assessed using an appropiate scale before insertion of the catheter, during the procedure and after removal of catheter
Patients degree of breathlessnesss (score) | from date of indication until removal of catheter, assessed up until 3 month
  Breathlessness will be assessed using an appropiate scale before insertion of the catheter, during the procedure and after removal of catheter
Patients satisfaction | On the date of removal, assessed up until 1 month
  After removal of catheter patients will be given a questionnaire
72- hour revisit from discharged (count) | from date of discharge and up until 72 hours
  Defined as any unplanned hospital stay within 72 hours from previous hospital discharge
30 days re-admission (count) | from date of discharge and up assessed until 30 days
  defined as any admission during 30 day follow-up
Complications to thoracentesis (count) | from insertion of catheter and assessed up until 1 week after removal of catheter
  Number of complications to thoracentesis
Total ED admission time (days) | From date and time for admission until date and time for ED discharge, assessed up until 1 month
  Date and time for admission until date and time for ED discharge
Total volume drained ( ml) | from date of insertion of catheter until removal of catheter, assessed up until 3 month
  the total amount of fluid drained from insertion of catether until removal of cathether

CONTACTS AND LOCATIONS:
Overall Officials: Sandra T Langsted, Principal Investigator — Aarhus University Hospital
Locations (6):
- Denmark (6):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Gødstrup Regional Hospital, Gødstrup, Central Jutland
  - Horsens Regional Hospital, Horsens, Central Jutland
  - Randers Regional Hospital, Randers, Central Jutland
  - Aalborg University Hospital, Aalborg, North Denmark
  - Esbjerg sygehus, Esbjerg, South Region Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified data necessary to reproduce published results will be made available on reasonable requests.
Time Frame: Six months after the publication of the last results, all de-identified individual patient data will be made available upon request. There will be no predetermined end date for the data sharing.